CLINICAL TRIAL: NCT04377581
Title: COVID-19 Health Messaging Efficacy and Its Impact on Public Perception, Anxiety, and Behavior
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: The Huck Institutes of the Life Sciences (Unknown); The Social Science Research Institute (Unknown); The Department of Family and Community Medicine, Penn State College of Medicine (Unknown); The College of Healthcare Information Management Executives (CHIME) (Unknown)
Responsible Party: Principal Investigator, Robert Lennon, Associate Professor, Family and Community Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY00014798
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Public Health; Demography; Pandemics; Corona Virus Infection; News; Global Health; Perception
Keywords: Penn State; CHIME; COVID-19 Messaging Study
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Effective communication is a critical component of managing pandemic outbreaks like COVID-19. This study explores COVID-19 related public knowledge, perceptions, belief in public health recommendations, intent to comply with public health recommendations, trust in information sources and preferred information sources. Participants are invited to include detailed free-text answers to make sure their COVID-19 experiences are heard.

DETAILED DESCRIPTION:
The survey is available online in 23 languages. Free-text responses in native languages are highly encouraged. A robust global response will not only provide invaluable information to inform clinicians, healthcare institutions and governments about how to optimize the content and venue of COVID-19 messaging, but will help write a Story of COVID in the words and languages of people from all over the world.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age

Exclusion Criteria:

* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Human Adults
Sampling Method: Non-Probability Sample
Enrollment: 18251 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Knowledge and Confidence in Knowledge of COVID-19 | Through study completion, an average of 3 months.
  Binary knowledge measures (true/false questions pertaining to COVID-19) each have a corresponding 5-point confidence score, the inverse of which generates a weighting variable. Weighted knowledge scores will be analyzed via a generalized linear mixed-methods effects model with a logistic link function and a random effect for the participant, generating a probability of correct response from 0 to 1.0.
Beliefs about the effectiveness of public health recommendations | Through study completion, an average of 3 months.
  Participants are asked, "Do you think that following these CDC recommendations will decrease the spread of COVID-19 in your community?" and select from a 5-point scale, Minimum: 1=certainly not; Maximum: 5 = most certainly.
Intent to comply with public health recommendations | Through study completion, an average of 3 months.
  Participants are asked, "Will you follow these recommendations?" and select from a 5-point scale, Minimum: 1=certainly not; Maximum: 5 = most certainly.
Perception of Risk of COVID-19 and other health threats | Through study completion, an average of 3 months.
  Participants are asked, "How likely is it that you will be diagnosed with any of the following diseases over the next year?" and rate their perceived likelihood of diagnosis for Measles, Flu, Lung Cancer, Ebola and COVID-19 on a 5 point scale. Minimum: 1, very unlikely; Maximum: 5, very likely.
  Participants are asked, "How serious do you think infection with any of the following diseases would be (or is) to your own personal health?" and rate their perceived seriousness of diagnosis for Measles, Flu, Lung Cancer, Ebola and COVID-19 on a 5 point scale. Minimum: 1, Not at all Serious; Maximum: 5, Very Serious
Perceptions of trust in common health information sources | Through study completion, an average of 3 months.
  Participants are asked the extent to which they trust common information sources: The World Health Organization, The U.S. Centers for Disease Control and Prevention, the European Commission, the participant's national government, the participant's local government, and the participant's personal healthcare provider. Participants rate on a 5 point scale. Minimum: 1, Not at all; Maximum: 2, Completely. (As these sources are not recognized in all places, participants may select "Not Applicable" in lieu of ranking.
Single most trusted news source | Through study completion, an average of 3 months.
  Participants are asked to identify their single most trusted source of news through selection from a pre-generated list or via free-text.

SECONDARY OUTCOMES:
Intention to change consumption of news because of COVID-19 (yes/no) | Through study completion, an average of 3 months.
  Participants are asked if COVID-19 will change how they consume news (y/n)
For participants who will change their news consumption, in what way will they change? | Through study completion, an average of 3 months.
  Participants who answer, "Yes" to Outcome 7 are asked to provide a free-text response to describe how their consumption of news will change.
Secondary information sources | Through study completion, an average of 3 months.
  Participants are asked to identify all other sources of information via selection from pre-generated menu or free-text.
Concerns about COVID-19 | Through study completion, an average of 3 months.
  Free-text response invited to describe their concerns regarding COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Lennon, MD, JD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States